CLINICAL TRIAL: NCT02721927
Title: The Use of Emergency Department by Syrian Refugees and the Increasing Cost of Health Care
Status: Completed | Type: Observational
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Umut Gulacti, Principal Investigator, Adiyaman University Research Hospital
Other Study IDs: ADYU 3
Record Dates: First submitted 2016-03-23; First posted 2016-03-29 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Emergency
Keywords: refugees; Syrian; cost; visit
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Syrian Refugees — Adult Syrian patients who visited the Emergency Department
  Other Names: Syrian Refugee patient

SUMMARY:
Since the beginning of the Syria conflict in March 2011, more than 10 million Syrians were forced to leave their homes and sought refuge in neighboring countries.

DETAILED DESCRIPTION:
Since the beginning of the Syria conflict in March 2011, more than 10 million Syrians were forced to leave their homes and sought refuge in neighboring countries (). In the result influx of the thousands of Syrian migrants who continue to cross into world, all the world especially the European countries faced with a huge refugee problem. Emergency medicine is play key role of being healthcare's safety net, being the last resort for those with no primary healthcare and no alternatives.

The aim of this study was to evaluate the use of Emergency Department by Syrian refugees and total and costs of their health care.

ELIGIBILITY:
Inclusion Criteria:

* Adult Syrian patients who visited the Emergency Department were included in the study.

Exclusion Criteria:

* Patients below 18 years of age
* Emergency Department returns during same day
* Patients with missing data in hospital medical record were excluded from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult Syrian patients who visited the Emergency Department of Adiyaman University of Training and Research Hospital between 1 January 2015 and 1 January 2016 retrospectively.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the use of Emergency department by Syrian refugees | one year
  Evaluate the emergency department visits of Syrian refugees by data obtained from hospital medical record

CONTACTS AND LOCATIONS:
Overall Officials: Umut Gulacti, Principal Investigator — Adiyaman University of Medical Faculty
Locations (1):
- Adiyaman University Research Hospital, Adıyaman, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Karakus A, Yengil E, Akkucuk S, Cevik C, Zeren C, Uruc V. The reflection of the Syrian civil war on the emergency department and assessment of hospital costs. Ulus Travma Acil Cerrahi Derg. 2013 Sep;19(5):429-33. doi: 10.5505/tjtes.2013.78910. PMID 24214784